CLINICAL TRIAL: NCT04912687
Title: Implementing Circulating Tumor DNA Analysis at Initial Diagnosis to Improve Management of Advanced Non-small Cell Lung Cancer Patients (NSCLC)
Brief Title: Implementing Circulating Tumor DNA Analysis at Initial Diagnosis to Improve Management of Advanced NSCLC Patients
Acronym: CIRCULAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IB 2021-02; 2021-A00685-36 (Other: ANSM IDRCB Number)
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer; Advanced Solid Tumor
Keywords: non-small cell lung cancer; EGFR detection; liquid biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This is a multicentric prospective cohort in which newly diagnosed advanced NSCLC patients will be included. For all patients, both tumor and liquid biopsy samples will be used for sequencing and detection of EGFR gene mutation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): For all patients, blood sample will be collected at inclusion (liquid biopsy) for sequencing.
  As per standard management, for all of these patients, EGFR gene mutation will be also analyzed on archived tumor sample.
  Interventions: Diagnostic Test: EGFR gene mutation analysis on liquid biopsy

INTERVENTIONS:
Diagnostic Test: EGFR gene mutation analysis on liquid biopsy — Blood samples will be collected at inclusion for plasma DNA collection and analysis.

SUMMARY:
Multicenter prospective cohort study aiming to evaluate the detection rate of EGFR gene mutation in patients with advanced NSCLC in a real-word clinical setting, based on liquid biopsy and tissue analyses.

DETAILED DESCRIPTION:
This a multicenter prospective cohort study. This study will be proposed to newly diagnosed advanced NSCLC patients. For included patients, archived paraffin embedded tumor tissue will be used for sequencing ; and blood sample will be collected for research purpose (plasma DNA collection and sequencing).

Both tissue and liquid biopsy samples will follow usual processes and will be sent to the Molecular Pathology laboratory of the Investigation center.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years at time of proposal study,
2. Histologically confirmed non-small cell lung carcinoma,
3. No previous treatment for NSCLC,
4. Indication to EGFR status determination following HAS recommendation,
5. Voluntary signed and dated written informed consent prior to any study specific procedure
6. Patients with a social security in compliance with the French Law.

Exclusion Criteria:

1. Treatment for advanced NSCLC started before liquid biopsy sampling.
2. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To assess the detection rate of patients with an EGFR actionable alteration when using the combination of two diagnostic procedures which include liquid biopsy analysis (by droplet digital PCR or allele specific PCR) and tissue analysis | within 3 weeks after signature of informed consent
  Resuls of each EGFR diagnostic procedure will be categorized as EGFR positive in case of the presence of an EGFR actionnable alteration ; as EGFR negative in case of the absence of an EGFR actionnable alteration ; or nor interpretable. A patient will be considered to have an EGFR actionable alteration if the mutation has been detected on the sequencing of tumor tissue OR if it has been detected on the liquid biopsy procedure

SECONDARY OUTCOMES:
The detection rate of patients with an EGFR actionable alteration based on the use of liquid biopsy analysis only | within 3 weeks after signature of informed consent
  A patient will be considered to have an EGFR actionable alteration (EGFR+) detected by the liquid biopsy analysis if an EGFR actionable alteration is identified based on the liquid biopsy analysis
The detection rate of patients with an EGFR actionable alteration based on tissue analysis only | within 3 weeks after signature of informed consent
  A patient will be considered to have an EGFR actionable alteration (EGFR+) detected by tissue analysis if an EGFR actionable alteration is identified based on the sequencing of tumor tissue
The concordance and discordance rates between the two procedures | within 3 weeks after signature of informed consent
  Concordance is defined whenever results of both techniques are identical (i.e. EGFR+ for both techniques or EGFR- for both techniques). Discordance is defined whenever results of both techniques are different.
The failure rate for each procedure and reasons of failure (insufficient DNA quantity, poor DNA quality, insufficient tissue quantity, poor tissue quality, analytical failure) | within 3 weeks after signature of informed consent
  •
  Failure of a procedure (sequencing of tumor tissue or liquid biopsy) is defined whenever the procedure fails to provide an interpretable result (Reasons for failure will be collected, i.e. insufficient DNA quantity, poor DNA quality, insufficient DNA/tissue quantity, poor DNA/tissue quality, analytical failure)
Delay to obtain sequencing results | within 3 weeks after signature of informed consent
  The delay between the date of the signature of the informed consent and the date of availability of the results for each procedure
Delay for treatment initiation | within 3 months after signature of informed consent
  The delay between the date of sample collection and the date of treatment initiation

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Institut Bergonie, Bordeaux
  - CHRU Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU Nice-Hopital de Cimiel, Nice
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - CHU de Rennes - Hopital Pontchaillou, Rennes
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No